CLINICAL TRIAL: NCT04938284
Title: The Synergistic Effect of Paired Associative Stimulation and Vagus Nerve Stimulation on Motor-evoked Potential Potentiation in Healthy Subjects
Brief Title: Combining PAS to Non-invasive VNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anastasia Shulga, Head of Department, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UAK1022001
Record Dates: First submitted 2021-06-11; First posted 2021-06-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Spinal Plasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PAS and VNS (Experimental)
  Interventions: Device: PAS; Device: VNS
- PAS and sham VNS (Active Comparator)
  Interventions: Device: PAS
- PAS (Active Comparator)
  Interventions: Device: PAS
- VNS (Active Comparator)
  Interventions: Device: VNS

INTERVENTIONS:
Device: PAS — Paired associative stimulation is a combination of non-invasive transcranial magnetic stimulation (TMS) and non-invasive peripheral nerve stimulation (PNS)
  Arms: PAS; PAS and VNS; PAS and sham VNS
Device: VNS — Non-invasive vagus nerve stimulation delivered through cymba concha & cymba cavum of the ear.
  Arms: PAS and VNS; VNS

SUMMARY:
Vagus nerve stimulation (VNS) and paired associative stimulation (PAS) have been shown to have efficacy in improving the results of motor rehabilitation after stroke and spinal cord injury, respectively. Here we will investigate in healthy subjects the synergistic effect of these stimulation modalities on motor-evoked potential (MEP) potentiation.

ELIGIBILITY:
Exclusion Criteria:

* contraindications to TMS (e.g. brain pathology, implanted devices)
* contraindications to MRI (e.g. MRI incompatible implants)
* continuous use of CNS-active drugs
* neurological, psychiatric or cardiovascular disease
* drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential (MEP) potentiation | 0 minutes after the stimulation protocol
  MEPs are responses to transcranial magnetic stimulation recorded from target muscles.
Motor evoked potential (MEP) potentiation | 30 minutes after the stimulation protocol
  MEPs are responses to transcranial magnetic stimulation recorded from target muscles.
Motor evoked potential (MEP) potentiation | 60 minutes after the stimulation protocol
  MEPs are responses to transcranial magnetic stimulation recorded from target muscles.
Motor evoked potential (MEP) potentiation | 90 minutes after the stimulation protocol
  MEPs are responses to transcranial magnetic stimulation recorded from target muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Background] Shulga A, Lioumis P, Kirveskari E, Savolainen S, Makela JP. A novel paired associative stimulation protocol with a high-frequency peripheral component: A review on results in spinal cord injury rehabilitation. Eur J Neurosci. 2021 May;53(9):3242-3257. doi: 10.1111/ejn.15191. Epub 2021 Mar 29. PMID 33738876
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- [Result] Haakana P, Natkynmaki A, Kirveskari E, Makela JP, Kilgard MP, Tarvainen MP, Shulga A. Effects of auricular vagus nerve stimulation and electrical earlobe stimulation on motor-evoked potential changes induced by paired associative stimulation. Eur J Neurosci. 2024 Oct;60(8):5949-5965. doi: 10.1111/ejn.16539. Epub 2024 Sep 11. PMID 39258329